CLINICAL TRIAL: NCT01295112
Title: Effect of Ozurdex® 0.7 mg on Improvement of Efficacy of Bevacizumab Therapy for Non-Ischemic Central Retinal Vein Occlusion
Brief Title: Effect of Ozurdex® 0.7 mg on Improvement of Efficacy of Bevacizumab for Central Retinal Vein Occlusion
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Texas Retina Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRA-OZAB-11-001
Record Dates: First submitted 2011-02-10; First posted 2011-02-14 (Estimated); Results first posted 2017-10-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2017-09

CONDITIONS: Non-Ischemic Central Retinal Vein Occlusion
MeSH Terms: interventions — Bevacizumab; Calcium Dobesilate; Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Sham Comparator): Active bevacizumab (Avastin®) and Sham Ozurdex®
  Interventions: Drug: Active bevacizumab and Sham dexamethasone
- Group 2 (Active Comparator): Active bevacizumab (Avastin®) and Active Ozurdex®
  Interventions: Drug: Active bevacizumab and Active dexamethasone

INTERVENTIONS:
Drug: Active bevacizumab and Sham dexamethasone — Bevacizumab: 25 mg/mL, PRN dosing Sham dexamethasone intravitreal implant: blunt needling of the sclera with no penetration of the globe
  Other Names: Avastin® (bevacizumab); Ozurdex® (dexamethasone intravitreal implant)
  Arms: Group 1
Drug: Active bevacizumab and Active dexamethasone — Bevacizumab: 25 mg/mL, PRN dosing Dexamethasone intravitreal implant: 0.7 mg, single dose
  Other Names: Avastin® (bevacizumab); Ozurdex® (dexamethasone intravitreal implant)
  Arms: Group 2

SUMMARY:
This is a study designed to determine if the addition of Ozurdex® to bevacizumab (Avastin®) eye injections reduces the need for repeat bevacizumab eye injections in patients with nonischemic central retina vein occlusion.

DETAILED DESCRIPTION:
This is a multicenter clinical study designed to determine if the addition of Ozurdex® injection to bevacizumab (Avastin®) eye injections reduces the need for repeat bevacizumab eye injections in patients with nonischemic central retina vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. male or female subjects (aged 18 or older);
2. provide written informed consent and sign/date a health information release;
3. women of childbearing potential must be willing to practice effective contraception for the duration of the study.

Exclusion Criteria:

1. any systemic disease or clinical evidence of any condition which would make the subject, in the opinion of the investigator, unsuitable for the study or could potentially confound the study results;
2. use of systemic steroids within 1 month prior to Baseline Visit (Visit 1) or anticipated use at any time during the study (inhaled and intranasal steroids are allowed);
3. sitting systolic blood pressure equal to or greater than 160 mmHg or diastolic blood pressure equal to or greater than 100 mmHg at the Baseline Visit (Visit 1);
4. use of warfarin, heparin, enoxaparin or similar anticoagulants within 2 weeks prior to Baseline Visit (Visit 1) or anticipated use at any time during the study;
5. known allergy or hypersensitivity to the study medications or their components;
6. previous enrollment in an Ozurdex® clinical trial or previous use of an Ozurdex® implant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Csaky, MD, Principal Investigator — Texas Retina Associates
Locations (1):
- Texas Retina Associates, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 68 participants ≥18 years of age with a diagnosis of central retinal vein occlusion (CRVO) as determined by fundus photography and fluorescein angiography were enrolled in the study at 5 clinical centers.
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 35 | 33
Completed | 35 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 35 | 33 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (15.0) | 70.7 (12.6) | 68.5 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 22 | 17 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black | 2 | 1 | 3
  Caucasian | 25 | 24 | 49
  Hispanic | 5 | 5 | 10
  Not Reported | 2 | 2 | 4
Previous Injections [Count of Participants; unit: Participants]
  Bevacizumab | 5 | 8 | 13
  No Injection | 22 | 21 | 43
  Ranibizumab | 4 | 3 | 7
  Bevacizumab and Ranibizumab | 1 | 1 | 2
  Bevacizumab and Aflibercept | 3 | 0 | 3
Study Eye [Count of Participants; unit: Participants]
  Right Eye | 18 | 15 | 33
  Left Eye | 17 | 18 | 35
Baseline best corrected visual acuity (BCVA) in Study Eye [Mean (Standard Deviation); unit: letters] — Best corrected visual acuity (BCVA): best possible vision a person can achieve with corrective lenses, measured using the method from the early treatment for diabetic retinopathy study (ETDRS) protocol. BCVA ranges from 0 to 100.
  letters | 49.6 (18.2) | 55.7 (17.2) | 52.5 (17.8)
Baselinen best corrected visual acuity (BCVA) in Fellow Eye [Mean (Standard Deviation); unit: letters] — Best corrected visual acuity (BCVA): best possible vision a person can achieve with corrective lenses, measured using the method from the early treatment for diabetic retinopathy study (ETDRS) protocol. BCVA ranges from 0 to 100.
  letters | 82.0 (12.6) | 82.2 (9.6) | 82.1 (11.2)
Baseline Central Foveal Thickness in Study Eye [Mean (Standard Deviation); unit: microns] | 264.5 (68.9) | 262.1 (70.0) | 263.3 (68.8)
Baseline Central Foveal Thickness in Fellow Eye [Mean (Standard Deviation); unit: microns] | 209.3 (39.1) | 213.1 (35.6) | 211.2 (36.9)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint is the Total Number of PRN Bevacizumab Intravitreal Injections Through 24 Weeks
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 35 | 33
Participants
  0 PRN Injections | 5 | 19
  1 PRN Injection | 13 | 11
  2 PRN Injections | 10 | 3
  3 PRN Injections | 6 | 0
  4 PRN Injections | 1 | 0
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority; p = 0.00002, Cochran-Mantel-Haenszel

2. Secondary Outcome: The Secondary Efficacy Endpoint is the Visual Acuity Score Based on Best Corrected Visual Acuity (BCVA) at Week 24
Description: The secondary efficacy endpoint is the visual acuity score based on best corrected visual acuity (BCVA) at Week 24 Change in BCVA at Week 24 from baseline
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 35 | 33
letters | 16.20 (15.49) | 13.55 (19.41)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Non-Inferiority — Non-inferiority will be described by the 95% upper bound of the confidence interval on the difference in the improvement from baseline in BCVA; p = 0.53, t-test, 1 sided — The p-value is assume superiority. The 95% upper confidence (upper end of the 90% Confidence interval) interval for the non-inferiority analysis is provided below; Mean Difference (Final Values) = 2.51, 90% CI 2-sided [-4.43 to 9.74], Standard Deviation 17.96

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/33
Other Adverse Events (participants affected / at risk) | 0/35 | 0/33

LIMITATIONS AND CAVEATS:
Limitations of this study included the relatively small size of 68 eyes, however statistical analyses were robust. The sample size was small due to the disease of study being a rare disease of study so the sample size is limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No